CLINICAL TRIAL: NCT06167356
Title: Observational Study on the Occurrence of Possible Relapses and on the Quality of Life in Patients Who Underwent Endoscopic Resection Surgery for Bladder Cancer (TURBK).
Brief Title: Study on the Occurrence of Possible Relapses and on the Quality of Life in Patients Who Underwent TURBK.
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Francesco Montorsi, Professor, IRCCS San Raffaele
Other Study IDs: Prot. 2007-Vescica
Record Dates: First submitted 2023-10-12; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Non Muscle Invasive Bladder Cancer; Non-Muscle Invasive Bladder Neoplasms; Non-Muscle Invasive Bladder Urothelial Carcinoma; Bladder Cancer; Bladder Disease; Bladder Neoplasm; Bladder Urothelial Carcinoma; Bladder Cancer Stage I, With Cancer in Situ; Bladder Cancer Recurrent; Bladder Urothelial Carcinoma in Situ; Bladder Urothelial Dysplasia
Keywords: Intravescical Therapies; Bladder Urothelial Carcinoma; Bladder Neoplasm; Bladder Disease; Bladder Cancer; Intravesical Instillations
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms; Urinary Bladder Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with non-muscle invasive bladder cancer: Patients with non-muscle invasive bladder cancer who underwent one of the following endoscopic resection surgeries : TURBK, MAPPING, TURBK SECOND LOOK, BLADDER BIOPSIES

SUMMARY:
A database has been created and will be used in which data will be collected in electronic format relating to adult patients who underwent one of the following endoscopic resection surgeries: TURBK, MAPPING, TURBK SECOND LOOK, BLADDER BIOPSIES.

DETAILED DESCRIPTION:
Each patient will be followed for approximately 10 years starting from the date of surgery. The patient may be contacted for yearly follow-up through one of the preferred methods indicated (phone call, email or home address) which will be carried out by the staff of the Urology Department. The data for each patient will then be transferred to the database itself. The data collected will be handled follwing the most strict GCPs and privacy norms.

The data entered will concern:

* period before hospitalization (symptoms, clinical data) and completion of a pre-surgery questionnaire
* hospitalization period with all its related data
* questionnaires relating to quality of life which will be administered to the patient once a year according to the preferred method expressed by the patient in the informed consent.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Patients with non-muscle invasive bladder cancer
* Indication to cancer removal through endoscopic resection surgery
* Ability to read and sign the informed consent

Exclusion Criteria:

* Age <18 years
* Inability to read and sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non muscle-invasive bladder cancer who underwent one of the following endoscopic resection surgeries : TURBK, MAPPING, TURBK SECOND LOOK, BLADDER BIOPSIES
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2013-11-27 (Actual); Primary Completion 2063-11-27 (Estimated); Study Completion 2063-11-27 (Estimated)

PRIMARY OUTCOMES:
obtain health benefit for the patients themselves and for future patients suffering from bladder cancer | 1 Annual follow-up from the date of surgery until the date in which patient decides to stop providing follow-up responses or until the date of death from any cause.
  All patients, before underwent endoscopic resection surgery, receive a diary in which we ask a detailed clinical history of the patient with their symptoms, diagnosis and previous urological e non urological treatments performed before the operation. A detailed intraoperative, postoperative and follow-up clinical history
improve the patient's scientific knowledge and develop new procedures for the diagnosis and treatment of the patient | 1 Annual follow-up from the date of surgery untile the date in which patient decides to stop providing follow-up responses or until the date of death from any cause.
  Through the collection of a detailed clinical history of the patient in which themselves report symptoms, diagnosis and previous urological and non-urological treatments and also through the medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Montorsi, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No